CLINICAL TRIAL: NCT01526018
Title: The Bottle Study: Infant Weight Gain During Use of Novel Versus Typical Infant Feeding Bottles
Status: Terminated | Type: Observational
Why Stopped: Inadequate recruitment
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Paula Chandler-Laney, PhD, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: F110921001
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Infant Feeding Behavior
Keywords: Intake; Formula feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Novel bottle
  Interventions: Behavioral: Podee bottle

INTERVENTIONS:
Behavioral: Podee bottle — Infants will acclimate to the Podee bottle over the course of several weeks. All infants will consume meals from the Podee and their usual bottles.

SUMMARY:
The purpose of this study is to pilot test whether a novel infant feeding bottle changes how much formula an infant drinks and how quickly he/she drinks it, as compared to meals provided in a standard bottle. Exclusively formula-fed infants and their caregiver will be provided with the novel feeding bottle and caregivers will be asked to acclimate their infant to this bottle during the next several weeks. Once acclimated, infants will undergo two weighed, timed, and videotaped test meals on two separate days; one with the novel bottle and one with their standard bottle, in random order. It is hypothesized that when the novel bottle is used, infants bottle will consume smaller meals and will have a longer meal duration, as compared to when a standard bottle is used.

ELIGIBILITY:
Inclusion Criteria:

* healthy, exclusively formula-fed infants aged 1-6 months at enrollment;
* parent must be at least 19 years of age, able to understand written and verbal English, and provide daytime care for the infant at least 4 days per week.

Exclusion Criteria:

* born < 37 weeks;
* birth weight < 2500g or > 4000g;
* current weight < 10th percentile for age;
* hospitalization > 72 hours following birth or any hospital admission since birth;
* any health issue that could interfere with feeding and/or growth;
* use of complementary foods;
* inability or unwillingness to comply with study-related procedures.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Bottle-fed infants aged 1-6 months
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Food intake | 2 weeks
  Rate of intake, volume of intake, duration of meal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States